CLINICAL TRIAL: NCT02881853
Title: Safety, Tolerability, and Bioavailability of Subcutaneously Administered XmAb®7195
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Collaborators: ICON Early Phase Services, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: XmAb7195-02
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Healthy Volunteers; Atopic Disease
Keywords: healthy; atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Part A1 (Experimental): XmAb7195 for IV infusion; dose level 1; 4 once-weekly doses
  Interventions: Drug: XmAb7195
- Part A2 (Experimental): XmAb7195 for SC injection; dose level 1; 4 once weekly doses
  Interventions: Drug: XmAb7195
- Part A3 (Experimental): XmAb7195 for SC injection; dose level 2; 4 once weekly doses
  Interventions: Drug: XmAb7195
- Part A4 (Experimental): XmAb7195 for SC injection; dose level 3; 4 once weekly doses
  Interventions: Drug: XmAb7195
- Part A5 (Experimental): XmAb7195 for SC injection; dose level 4; 4 once weekly doses
  Interventions: Drug: XmAb7195
- Part B6 (Experimental): XmAb7195 or placebo for SC injection; dose level 5; 4 once-weekly doses
  Interventions: Drug: XmAb7195; Drug: Placebo
- Part B7 (Experimental): XmAb7195 or placebo for SC injection; dose level 6; 4 once-weekly doses
  Interventions: Drug: XmAb7195; Drug: Placebo
- Part B8 (Experimental): XmAb7195 or placebo for SC injection; dose level 7; 4 once-weekly doses
  Interventions: Drug: XmAb7195; Drug: Placebo
- Part B9 (Experimental): XmAb7195 or placebo for SC injection dose level 8; 4 once-weekly doses
  Interventions: Drug: XmAb7195; Drug: Placebo

INTERVENTIONS:
Drug: XmAb7195
Drug: Placebo
  Arms: Part B6; Part B7; Part B8; Part B9

SUMMARY:
This is a Phase 1b, combined multiple dose subcutaneous (SC) bioavailability (BA) and multiple ascending dose (MAD) study evaluating safety, tolerability and BA of SC XmAb7195 in healthy subjects and in subjects with atopic disease.

DETAILED DESCRIPTION:
The study will be divided into 2 parts. Part A will be an open-label, parallel group, BA study evaluating 4 once-weekly doses of IV XmAb7195 or SC XmAb7195 in healthy subjects. Each of 5 treatment groups will consist of 6 subjects. Part B will commence following the completion of Part A and will be a randomized, double-blind, placebo-controlled, MAD study evaluating 4 once weekly doses of SC XmAb7195 in healthy subjects and/or subjects with atopic disease. Each treatment group will consist of 8 subjects randomized 3:1 to XmAb7195:placebo Subjects in both parts of the study will be followed for at least 28 days after their last dose.

ELIGIBILITY:
Inclusion Criteria:

All Subjects:

* Male or female between 18 to 60 years of age (inclusive at the time of screening).
* Total body weight 50.0 to 100.0 kg, and body mass index (BMI) 19.0 to 35.0 kg/m2 (inclusive, at screening).
* Women can be of either childbearing or non-childbearing potential.
* Must be healthy with no clinically significant abnormality identified on medical or laboratory evaluation and no history of any clinically significant disorder, condition, or disease that would pose a risk to subject or interfere with the study evaluation, procedures, or completion as assessed by the Investigator.

Subjects with Atopic Disease Only (Part B):

* Allergen skin test reactivity of ≥ 5 mm wheal greater than saline control to any 2 of the following 5 allergens: D. pteronyssinus, D. farina, ragweed, Virginia live oak, and mountain cedar within 21 days prior to dosing.
* Sufficient clinical control of subject's atopic disease such that, in the opinion of the Investigator, the subject is unlikely to require substantial changes in therapy medication for the duration of the trial and unlikely to require the addition of an exclusionary medication

Exclusion Criteria:

* Subjects who have a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases, or disorders that would pose a significant risk to subject's safety or significantly interfere with the study evaluation, procedures, or completion as assessed by the Investigator.
* Subjects with platelet count < 150 k/uL at screening or at the time of initial admission.
* Subjects with peak expiratory flow rate < 400 L/min for males and < 350 L/min for females.
* Subjects with conditions associated with high risk of bleeding such as: past history of intracranial or gastrointestinal bleeding, hemorrhagic condition including hereditary or acquired bleeding, or coagulation disorder.
* Subjects with history of any clinically significant cardiovascular event such as: myocardial infarction, acute coronary syndrome, stroke, pulmonary embolism, and/or deep venous thrombosis.
* Subjects who do not agree to use medically acceptable methods of contraception (as defined in the protocol).
* Subjects who are pregnant or breast feeding, or planning to become pregnant within 30 days of last dose of XmAb7195.
* Subjects who have used prescription drugs within 28 days prior to randomization with the following exceptions for Part B subjects with atopic disease:

  1. Intranasal corticosteroids for allergic symptoms if the dose has been stable for 14 days prior to randomization.
  2. Inhaled short acting beta agonist (SABA) therapy for bronchospasm if dosing has been stable for 14 days prior to randomization.
  3. No other prescription drugs are allowed unless agreed as not clinically relevant by the Investigator and Sponsor.
* Subjects who have had an asthma exacerbation requiring hospitalization within the 1 year prior to randomization or having required oral corticosteroids within the 6 months prior to randomization.
* Subjects with poorly controlled asthma defined as SABA > 6 times/day on any day within the 4 weeks prior to randomization.
* Subjects who have used any of the following medications within the 3 months prior to randomization: oral or inhaled corticosteroids, long acting beta agonists (LABAs), leukotriene receptor antagonists (LTRAs), or any other asthma controller medication (occasional SABA use is allowed).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-02-24 (Actual)

PRIMARY OUTCOMES:
Bioavailability of SC XmAb7195 after 4 once-weekly doses as measured by the ratio of dose-normalized SC XmAb7195 area under the concentration-time curve (AUC) to dose-normalized IV XmAb7195 AUC. | Date of randomization up to Day 50

SECONDARY OUTCOMES:
Cmax, Maximum observed serum concentration | Date of randomization up to Day 50
Time at which Cmax was observed [Tmax] | Date of randomization up to Day 50
Area Under the Curve (AUC) | Date of randomization up to Day 50
Terminal elimination half-life [t1/2] | Date of randomization up to Day 50
Total body or systemic clearance [CL] | Date of randomization up to Day 50
Apparent volume of distribution at steady state [Vss] | Date of randomization up to Day 50
Immunogenicity of SC XmAb7195 and IV XmAb7195 as measured by incidence of development of anti-XmAb7195 antibody after 4 once-weekly doses | Date of randomization up to Day 50

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel P DeNoia, MD, Principal Investigator — ICON Early Phase Services, LLC
Locations (1):
- ICON Early Phase Services, LLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No